CLINICAL TRIAL: NCT03404648
Title: Staging of Untreated Patients With Very High-risk and High-risk Prostate Carcinoma Utilizing Hybrid C11-choline PET/MR and Pelvic Multiparametric MRI for Personalized Precise Treatment: a Pilot Study
Brief Title: Staging Prostate Cancer With Hybrid C11-Choline PET/MR and mpMRI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ming Yang, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-007897
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Prostate Adenocarcinoma
Keywords: high risk; prostate cancer; C11-choline; PET/MR; mpMRI
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- High Risk Prostate Cancer Patients (Experimental): Subjects will receive C-11 choline PET Tracer and Gadobutrol prior to the one time Positron emission tomography (PET/MR scanner) imaging and Multiparametric Magnetic resonance imaging (mpMRI).
  Interventions: Drug: C-11 choline PET tracer; Drug: Gadobutrol; Device: PET/MR scanner

INTERVENTIONS:
Drug: C-11 choline PET tracer — C-11 choline PET tracer, One dose, totally 12-14 millicurie (mCi), intravenous administration while patient is lying on the table.
  Other Names: Choline C-11 Injection
Drug: Gadobutrol — Single dose of Gadavist® (Gadobutrol, Bayer) at no more than 0.1 mmol/kg will be administrated intravenously.
  Other Names: Gadavist
Device: PET/MR scanner — C11-PET/MR and pelvic mpMRI scan for prostate cancer.
  Other Names: GE SIGNA 3T PET/MR scanner

SUMMARY:
The purpose of this study is to find out if a PET/MR scan in combination with standard MRI and CT scans can improve the early detection and treatment of patients with prostate cancer.

DETAILED DESCRIPTION:
High risk prostate cancer patients will undergo C11-Choline PET/MR whole body fusion scan and pelvic mpMRI for accurate staging. The PET/MR imaging findings, including the primary lesion with the prostate bed and pelvic lymph nodes, will be correlated with the histopathologic result. Researchers aim to provide accurate one-stop shopping opportunity in diagnosis and staging of high risk prostate cancer using the C11-choline PET/MR scan.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated patients with high-risk and very high-risk prostate cancer, who require clinical pelvic mpMRI, CT, and bone scan as standard clinical care for diagnosis and management of prostate cancer.

Exclusion Criteria:

1. Patients who already received primary treatment or neo-adjuvant therapy.
2. Patients who refuse undergoing routine clinical imaging (i.e., pelvic mpMRI, CT, bone scan) for staging. Reimbursement of pelvic mpMRI in this study is denied. CT and bone scan may be done elsewhere outside of Mayo Clinic but should be of diagnostic quality. Research C-11 choline PET/MR will not substitute pelvic mpMRI, CT, or bone scan in this study.
3. Patients cannot tolerate MRI (e.g., claustrophobia, severe back pain or spasm, involuntary movement [e.g., tremor, dystonia]).
4. Patients have total hip arthroplasty (THA), which can cause substantial susceptibility artifact and degrade image quality of mpMRI.
5. Patients have cardiac pacemaker, cochlear implants, neurostimulator, medical device which is unsafe at 3 Tesla, or foreign metallic body in the eyes or orbit.
6. Patients have contraindication to gadolinium based MR contrast agents (e.g., renal failure, severe reaction to gadolinium based MR contrast agents). Epidermal growth factor receptor (eGFR) should be above 30 within 30 days the time of mpMRI.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ming Yang, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Risk Prostate Cancer Patients
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | High Risk Prostate Cancer Patients
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Uptake Value of C11-choline
Description: Measured by maximum standardized uptake value (SUVmax) of indexed lesions. SUV is calculated as ratio of concentration of tissue reactivity divided by dose at time of injection divided by body weight.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | High Risk Prostate Cancer Patients
Number analyzed (Participants) | 19
Ratio | 6.2 (1.8)

2. Primary Outcome: Number of Lesions Showing C11-Choline Uptake
Description: Measured by the mean number of lesions to show C11-Choline uptake.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | High Risk Prostate Cancer Patients
Number analyzed (Participants) | 19
Lesions | 1.2 (0.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 2 days on all participants.
Arm/Group | High Risk Prostate Cancer Patients
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT03404648/Prot_SAP_000.pdf